CLINICAL TRIAL: NCT03351738
Title: A Phase 2a Randomized, Double-blind, Placebo-controlled, Parallel-designed Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamic Effects of MEDI5884 in Subjects With Stable Coronary Heart Disease
Brief Title: A Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamic Effects of MEDI5884 in Adults With Stable Coronary Heart Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D7870C00002
Record Dates: First submitted 2017-10-12; First posted 2017-11-24 (Actual); Results first posted 2019-12-19 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Stable Coronary Heart Disease
Keywords: Coronary heart disease; Pharmacokinetic; Pharmacodynamics
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Placebo (Placebo Comparator): Participants will receive subcutaneous (SC) dose of placebo (volume matched to MEDI5884) on Days 1, 31, and 61.
  Interventions: Drug: Placebo
- MEDI5884 50 mg (Experimental): Participants will receive SC dose of MEDI5884 50 mg on Days 1, 31, and 61.
  Interventions: Drug: MEDI5884
- MEDI5884 100 mg (Experimental): Participants will receive SC dose of MEDI5884 100 mg on Days 1, 31, and 61.
  Interventions: Drug: MEDI5884
- MEDI5884 200 mg (Experimental): Participants will receive SC dose of MEDI5884 200 mg on Days 1, 31, and 61.
  Interventions: Drug: MEDI5884
- MEDI5884 350 mg (Experimental): Participants will receive SC dose of MEDI5884 350 mg on Days 1, 31, and 61.
  Interventions: Drug: MEDI5884
- MEDI5884 500 mg (Experimental): Participants will receive SC dose of MEDI5884 500 mg on Days 1, 31, and 61.
  Interventions: Drug: MEDI5884

INTERVENTIONS:
Drug: MEDI5884 — Participants will receive SC dose of MEDI5884 50 mg or 100 mg or 200 mg or 350 mg or 500 mg on Days 1, 31, and 61.
  Arms: MEDI5884 100 mg; MEDI5884 200 mg; MEDI5884 350 mg; MEDI5884 50 mg; MEDI5884 500 mg
Drug: Placebo — Participants will receive SC dose of placebo (volume matched to MEDI5884) on Days 1, 31, and 61.
  Arms: Placebo

SUMMARY:
A Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamic Effects of MEDI5884 in Adults With Stable Coronary Heart Disease.

DETAILED DESCRIPTION:
A Randomized, Double-blind, Placebo-controlled, Parallel-designed Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamic Effects of MEDI5884 in Participants with Stable Coronary Heart Disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stable coronary heart disease prior to screening
* Currently receiving high intensity statin(s)

Exclusion Criteria:

* Unstable cardiovascular conditions
* Any planned arterial revascularizations
* Fasting Laboratory values at screening: Triglycerides > 500 mg/dl, Low Density Lipoprotein-Cholesterol > 100 mg/dL
* Any disease or condition or laboratory value that would place the participant at an unacceptable risk.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2017-12-13 (Actual); Primary Completion 2018-11-09 (Actual); Study Completion 2018-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Koren, MD, FACC, Principal Investigator — Jacksonville Center For Clinical Research
Locations (23):
- United States (23):
  - Research Site, Anniston, Alabama
  - Research Site, Huntsville, Alabama
  - Research Site, El Cajon, California
  - Research Site, Lincoln, California
  - Research Site, Northridge, California
  - Research Site, Waterbury, Connecticut
  - Research Site, Fleming Island, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Pembroke Pines, Florida
  - Research Site, Port Orange, Florida
  - Research Site, Savannah, Georgia
  - Research Site, Evanston, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Louisville, Kentucky
  - Research Site, Fargo, North Dakota
  - Research Site, Cincinnati, Ohio
  - Research Site, Marion, Ohio
  - Research Site, Stow, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Rapid City, South Dakota
  - Research Site, Kingsport, Tennessee
  - Research Site, McAllen, Texas
  - Research Site, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ruff CT, Koren MJ, Grimsby J, Rosenbaum AI, Tu X, Karathanasis SK, Falloon J, Hsia J, Guan Y, Conway J, Tsai LF, Hummer BT, Hirshberg B, Kuder JF, Murphy SA, George RT, Sabatine MS. LEGACY: Phase 2a Trial to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamic Effects of the Anti-EL (Endothelial Lipase) Antibody MEDI5884 in Patients With Stable Coronary Artery Disease. Arterioscler Thromb Vasc Biol. 2021 Dec;41(12):3005-3014. doi: 10.1161/ATVBAHA.120.315757. Epub 2021 Oct 28. PMID 34706556
- See also: D7870C00002 Clinical Protocol Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D7870C00002&attachmentIdentifier=f8ee7185-f701-44eb-8222-5a66f56de14d&fileName=D7870C00002-protocol-amendment-4_redacted_2dec2019_FINAL.pdf&versionIdentifier=
- See also: D7870C00002 Statistical Analysis Plan Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D7870C00002&attachmentIdentifier=cd9a6d81-132c-42ac-850f-5371d1504545&fileName=D7870C00002_SAP_Redacted_21nov2019_FINAL.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in the US between 13Dec2017 and 09Nov2018.
Pre-assignment Details: A total of 248 participants consented to participate in the study, of which 115 were screen failures. A total of 133 participants were randomized to the study of which only 132 received treatment. One participant was ineligible, being randomized by error but not followed or treated.
Groups:
- Placebo: Participants received subcutaneous (SC) dose of placebo (volume matched to MEDI5884) on Days 1, 31, and 61.
- MEDI5884 50 mg: Participants received SC dose of MEDI5884 50 mg on Days 1, 31, and 61.
- MEDI5884 100 mg: Participants received SC dose of MEDI5884 100 mg on Days 1, 31, and 61.
- MEDI5884 200 mg: Participants received SC dose of MEDI5884 200 mg on Days 1, 31, and 61.
- MEDI5884 350 mg: Participants received SC dose of MEDI5884 350 mg on Days 1, 31, and 61.
- MEDI5884 500 mg: Participants received SC dose of MEDI5884 500 mg on Days 1, 31, and 61.
Period: Overall Study
Arm/Group | Placebo | MEDI5884 50 mg | MEDI5884 100 mg | MEDI5884 200 mg | MEDI5884 350 mg | MEDI5884 500 mg
Started | 23 | 20 | 24 | 22 | 21 | 22
Completed | 23 | 19 | 24 | 21 | 21 | 22
Not Completed | 0 | 1 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: As-treated population included all participants who received any dose of study drug and analyzed according to the treatment they actually received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | MEDI5884 50 mg | MEDI5884 100 mg | MEDI5884 200 mg | MEDI5884 350 mg | MEDI5884 500 mg | Total
Number analyzed (Participants) | 23 | 20 | 24 | 22 | 21 | 22 | 132
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.3 (8.4) | 63.8 (8.4) | 67.4 (5.7) | 64.7 (8.9) | 67.5 (7.8) | 67.6 (8.6) | 66.3 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 1 | 4 | 1 | 4 | 17
  Male | 19 | 17 | 23 | 18 | 20 | 18 | 115
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 2 | 0 | 1 | 1 | 7
  Not Hispanic or Latino | 21 | 19 | 22 | 22 | 20 | 21 | 125
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 0 | 0 | 0 | 0 | 2
  Black or African American | 1 | 1 | 1 | 2 | 1 | 2 | 8
  White | 21 | 17 | 23 | 20 | 20 | 19 | 120
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. The TEAEs are defined as events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug.
Time Frame: Day 1 (Baseline) through Day 241
Population: As-treated population: All participants who received any dose of study drug and analyzed according to actual treatment they received. Reported data are through Day 151 for all participants, and Day 241 for participants with elevated anti-drug antibodies (ADA), low-density lipoprotein cholesterol (LDL-C), triglycerides (TG) levels at Day 151 visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI5884 50 mg | MEDI5884 100 mg | MEDI5884 200 mg | MEDI5884 350 mg | MEDI5884 500 mg
Number analyzed (Participants) | 23 | 20 | 24 | 22 | 21 | 22
Participants
  TEAEs | 17 | 10 | 11 | 12 | 13 | 13
  TESAEs | 2 | 2 | 1 | 0 | 4 | 0

2. Primary Outcome: Number of Participants With Clinically Important Changes in Electrocardiograms (ECGs) From Baseline
Description: Number of participants with clinically important changes in ECGs from baseline are reported. Clinically important changes in ECGs is defined as any clinical significant difference in heart rate, RR interval, PR interval, QRS, and QT intervals from the primary lead of the digital 12-lead ECG from baseline.
Time Frame: Day 1 (Baseline) through Day 241
Population: As-treated population included all participants who received any dose of study drug and analyzed according to the treatment they actually received. Reported data are through Day 151 for all participants, and Day 241 for participants with elevated ADA, LDL-C, and TG levels at Day 151 visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI5884 50 mg | MEDI5884 100 mg | MEDI5884 200 mg | MEDI5884 350 mg | MEDI5884 500 mg
Number analyzed (Participants) | 23 | 20 | 24 | 22 | 21 | 22
Participants | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Clinically Important Changes in Vital Signs From Baseline
Description: Number of participants with clinically important changes in vital signs from baseline are reported. Vital signs measurements were obtained after the participant had rested in the supine position for at least 10 minutes at the recording time. Clinically important changes in vital signs from baseline is defined as any clinical significant difference in the vital sign parameters (blood pressure, heart rate, body temperature, and respiratory rate) from baseline.
Time Frame: Day 1 (Baseline) through Day 241
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI5884 50 mg | MEDI5884 100 mg | MEDI5884 200 mg | MEDI5884 350 mg | MEDI5884 500 mg
Number analyzed (Participants) | 23 | 20 | 24 | 22 | 21 | 22
Participants | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Clinically Important Changes in Laboratory Parameters From Baseline
Description: Number of participants with clinically important changes in laboratory parameters from baseline are reported. Clinically important changes in laboratory parameters is defined as any clinical significant difference in analysis of serum chemistry, hematology, and urine from baseline.
Time Frame: Day 1 (Baseline) through Day 241
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI5884 50 mg | MEDI5884 100 mg | MEDI5884 200 mg | MEDI5884 350 mg | MEDI5884 500 mg
Number analyzed (Participants) | 23 | 20 | 24 | 22 | 21 | 22
Participants | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Clinically Important Changes in Physical Examinations From Baseline
Description: Number of participants with clinically important changes in physical examinations from baseline are reported. Clinically important changes in physical examinations is defined as any clinical significant difference in general appearance, head, ears, eyes, nose, throat, neck, skin, heart, lung, abdomen, musculoskeletal system, endocrine system, nervous system, height, and weight from baseline.
Time Frame: Day 1 (Baseline) through Day 241
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI5884 50 mg | MEDI5884 100 mg | MEDI5884 200 mg | MEDI5884 350 mg | MEDI5884 500 mg
Number analyzed (Participants) | 23 | 20 | 24 | 22 | 21 | 22
Participants | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Change From Baseline in Apolipoprotein B
Description: Change from baseline in apolipoprotein B is reported.
Time Frame: Day 1 (Baseline), and Days 31, 61, and 91
Population: As-treated population included all participants who received any dose of study drug and analyzed according to the treatment they actually received. Here, "number analyzed" signifies number of participants analyzed for the specified time point.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | MEDI5884 50 mg | MEDI5884 100 mg | MEDI5884 200 mg | MEDI5884 350 mg | MEDI5884 500 mg
Number analyzed (Participants) | 23 | 20 | 24 | 22 | 21 | 22
mg/dL
  Day 31: number analyzed (Participants) | 23 | 19 | 24 | 22 | 21 | 21
  Day 31 | 3.3 (8.5) | 0.5 (12.2) | 5.1 (10.6) | 2.2 (9.4) | 7.1 (10.6) | 7.1 (14.3)
  Day 61: number analyzed (Participants) | 18 | 17 | 20 | 18 | 18 | 18
  Day 61 | 1.2 (13.9) | -1.2 (14.1) | 3.5 (10.8) | 2.6 (15.3) | 3.7 (11.7) | 6.2 (9.6)
  Day 91: number analyzed (Participants) | 21 | 19 | 24 | 21 | 21 | 22
  Day 91 | -0.5 (10.7) | 3.6 (29.3) | 2.3 (10.7) | 2.0 (8.3) | 2.9 (9.4) | 7.8 (13.4)

7. Secondary Outcome: Percent Change From Baseline in High Density Lipoprotein Cholesterol (HDL-C)
Description: Percent change from baseline in HDL-C is reported.
Time Frame: Day 1 (Baseline), and Days 31, 61, and 91
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Placebo | MEDI5884 50 mg | MEDI5884 100 mg | MEDI5884 200 mg | MEDI5884 350 mg | MEDI5884 500 mg
Number analyzed (Participants) | 23 | 20 | 24 | 22 | 21 | 22
Percent change
  Day 31: number analyzed (Participants) | 23 | 19 | 24 | 22 | 21 | 21
  Day 31 | -3.08 (10.28) | 7.37 (13.52) | 22.95 (25.04) | 27.25 (19.37) | 44.12 (24.74) | 55.80 (25.97)
  Day 61: number analyzed (Participants) | 18 | 17 | 20 | 18 | 18 | 18
  Day 61 | -4.69 (9.45) | 4.58 (12.45) | 28.28 (32.19) | 37.65 (22.76) | 39.74 (22.74) | 49.58 (21.46)
  Day 91: number analyzed (Participants) | 21 | 19 | 24 | 21 | 21 | 22
  Day 91 | -3.62 (13.41) | 1.98 (14.69) | 21.82 (30.66) | 35.63 (35.27) | 43.29 (31.09) | 48.31 (25.63)

8. Secondary Outcome: Area Under the Concentration-time Curve for 30 Days (AUC30d) After the Last Dose of MEDI5884
Description: AUC30d after the last dose of MEDI5884 is reported.
Time Frame: Day 61 (pre-dose), and on Days 64, 68, 71, and 91
Population: Pharmacokinetic (PK) evaluable population included all participants who received any dose of MEDI5884 with at least one detectable post treatment serum concentration measurement.
Measure: Mean (Standard Deviation); unit: μg⋅day/mL
Arm/Group | MEDI5884 50 mg | MEDI5884 100 mg | MEDI5884 200 mg | MEDI5884 350 mg | MEDI5884 500 mg
Number analyzed (Participants) | 18 | 22 | 20 | 20 | 20
μg⋅day/mL | 14.6 (27.3) | 51.8 (54.8) | 191 (176) | 584 (294) | 1020 (643)

9. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of MEDI5884 After the Last Dose
Description: Maximum observed serum concentration (Cmax) of MEDI5884 after the last dose is reported.
Time Frame: Day 61 (pre-dose), and on Days 64, 68, 71, 91, 111, and 151
Population: The PK evaluable population included all participants who received any dose of MEDI5884 with at least one detectable post treatment serum concentration measurement.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | MEDI5884 50 mg | MEDI5884 100 mg | MEDI5884 200 mg | MEDI5884 350 mg | MEDI5884 500 mg
Number analyzed (Participants) | 18 | 22 | 20 | 20 | 20
μg/mL | 1.01 (1.34) | 4.63 (2.95) | 11.9 (7.77) | 28.5 (13.0) | 46.3 (24.6)

10. Secondary Outcome: Terminal Elimination Half-life (t½) of MEDI5884 After the Last Dose
Description: Terminal half-life is the time required for the plasma concentration to fall by 50% during the terminal phase. The t½ of MEDI5884 after the last dose is reported.
Time Frame: Day 61 (pre-dose), and on Days 64, 68, 71, 91, 111, and 151
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | MEDI5884 50 mg | MEDI5884 100 mg | MEDI5884 200 mg | MEDI5884 350 mg | MEDI5884 500 mg
Number analyzed (Participants) | 0 | 2 | 7 | 14 | 14
Days |  | 7.56 (6.4) | 8.09 (2.80) | 10.3 (3.53) | 13.7 (5.86)

11. Secondary Outcome: Number of Participants With Treatment-emergent Anti-drug Antibodies (ADA) to MEDI5884
Description: Treatment-emergent ADA is defined as the sum of treatment-induced ADA (post baseline-positive only) and treatment-boosted ADA (baseline ADA titer that was boosted to a 4-fold or higher level following drug administration).
Time Frame: Day 1 (pre-dose), on Day 8, Day 31 (pre-dose), Day 61 (pre-dose), on Days 151 and 241
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI5884 50 mg | MEDI5884 100 mg | MEDI5884 200 mg | MEDI5884 350 mg | MEDI5884 500 mg
Number analyzed (Participants) | 23 | 20 | 24 | 22 | 21 | 22
Participants | 1 | 1 | 1 | 3 | 3 | 3

ADVERSE EVENTS:
Time Frame: Day 1 through Day 241
Arm/Group | Placebo | MEDI5884 50 mg | MEDI5884 100 mg | MEDI5884 200 mg | MEDI5884 350 mg | MEDI5884 500 mg
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/20 | 0/24 | 0/22 | 0/21 | 0/22
Serious Adverse Events (participants affected / at risk) | 2/23 | 2/20 | 1/24 | 0/22 | 4/21 | 0/22
Other Adverse Events (participants affected / at risk) | 9/23 | 9/20 | 6/24 | 12/22 | 13/21 | 13/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=23) | MEDI5884 50 mg (N=20) | MEDI5884 100 mg (N=24) | MEDI5884 200 mg (N=22) | MEDI5884 350 mg (N=21) | MEDI5884 500 mg (N=22)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral artery occlusion (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 4.3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=23) | MEDI5884 50 mg (N=20) | MEDI5884 100 mg (N=24) | MEDI5884 200 mg (N=22) | MEDI5884 350 mg (N=21) | MEDI5884 500 mg (N=22)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Vitreous adhesions (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Pancreatic cyst (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site bruising (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Injection site erythema (General disorders) | 2 (2) | 0 (0) | 1 (1) | 3 (5) | 4 (12) | 0 (0)
Injection site swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infected dermal cyst (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Apolipoprotein b increased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Blood triglycerides increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Crystal urine present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostatic specific antigen increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Calculus bladder (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Neurogenic bladder (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal cyst (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urine flow decreased (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nipple pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Allergic cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises on going studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-12-14): https://cdn.clinicaltrials.gov/large-docs/38/NCT03351738/SAP_001.pdf
  • Study Protocol (2018-05-29): https://cdn.clinicaltrials.gov/large-docs/38/NCT03351738/Prot_002.pdf